CLINICAL TRIAL: NCT02625324
Title: Valiant Evo International Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10219493DOC; NCT02625324 (Other: ClinicalTrials.gov)
Record Dates: First submitted 2015-12-02; First posted 2015-12-09 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Aortic Aneurysm, Thoracic
MeSH Terms: conditions — Aortic Aneurysm, Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Endovascular repair (Experimental): Valiant Evo Thoracic Stent Graft System
  Interventions: Device: Valiant Evo Thoracic Stent Graft System

INTERVENTIONS:
Device: Valiant Evo Thoracic Stent Graft System — Procedure: thoracic endovascular aneurysm repair (TEVAR)

SUMMARY:
The purpose of the Valiant Evo International Clinical Trial is to demonstrate the safety and effectiveness of the Valiant Evo Thoracic Stent Graft System in subjects with a descending thoracic aortic aneurysm (DTAA) who are candidates for endovascular repair.

DETAILED DESCRIPTION:
Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 total subjects, in order obtain 87 evaluable subjects for the primary endpoint. The two protocols are identical, and the trials were run simultaneously to enroll subjects concurrently in the United States (US) and Outside United States (OUS). The poolability on the primary endpoint between US and OUS data will be assessed using Fisher's exact test during the data analysis. Data for both trials will be combined and presented as a pooled analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years old
2. Subject understands and voluntarily has signed and dated the Patient Informed Consent approved by the Sponsor and by the Ethics Committee for this study
3. Subject presents a DTAA which is localized below the ostium of left subclavian artery (LSA) and above the ostium of celiac trunk
4. Subject has a DTAA that is one of the following:

   1. A fusiform aneurysm with a maximum diameter that:

      * is ≥ 50 mm and/or:
      * is ≥ 2 times the diameter of the non-aneurysmal thoracic aorta and/or:
      * is <50 mm and has grown ≥ 5 mm within previous 12 months
   2. A saccular aneurysm or a penetrating atherosclerotic ulcer
5. Subject's anatomy must meet all of the following anatomical criteria as demonstrated on contrast-enhanced CT and/or on contrast-enhanced MRI obtained within four (4) months prior to implant procedure:

   1. Proximal and distal non-aneurysmal aortic neck diameter measurements must be ≥ 16 mm and ≤ 42 mm
   2. Proximal non-aneurysmal aortic neck length must be ≥ 20 mm (for FreeFlo configuration) and ≥ 25 mm (for Closed Web configuration)
   3. Distal non-aneurysmal aortic neck length must be ≥ 20 mm
6. Subject has adequate arterial access site or can tolerate a conduit that allows endovascular access to the aneurysmal site with the delivery system of the appropriate sized device chosen for the treatment.

Exclusion Criteria:

1. Subject has a life expectancy of less than 1 year
2. Subject is participating in another investigational drug or device study which would interfere with the endpoints and follow-ups of this study
3. Subject is pregnant
4. Subject requires planned placement of the covered proximal end of the stent graft to occur in zones 0 or 1
5. Subject has a thoracic aneurysm with a contained rupture or localized at the anastomosis of a previous graft (pseudo-/false aneurysm)
6. Subject has a mycotic aneurysm
7. Subject has a dissection (type A or B) or an intramural hematoma or an aortic rupture in addition to the thoracic aneurysm
8. Subject requires emergent aneurysm treatment, e.g., trauma or rupture
9. Subject has received a previous stent or stent graft or previous surgical repair in the ascending and/or descending thoracic aorta, and/or in the aortic arch
10. Subject requires surgical or endovascular treatment of an infra-renal aneurysm at the time of implant
11. Subject has had previous surgical or endovascular treatment of an infra-renal aortic aneurysm
12. Treatment with the Valiant Evo Thoracic Stent Graft would require intentional revascularization of the brachio-cephalic artery, the left common carotid artery or the celiac trunk
13. Subject has had or plans to have a major surgical or interventional procedure within 30 days before or 30 days after the planned implantation of the Valiant Evo Thoracic Stent Graft. This does not include planned procedures that are needed for the safe and effective placement of the stent graft (i.e., carotid/subclavian transposition, carotid/subclavian bypass procedure)
14. Subject has a significant and/or circumferential aortic mural thrombus at either the proximal or distal attachment sites that could compromise fixation and seal of the implanted stent graft
15. Subject has a connective tissue disease (e.g., Marfan's syndrome, aortic medial degeneration)
16. Subject has a bleeding diathesis or coagulopathy, or refuses blood transfusion.
17. Subject has had a myocardial infarction (MI) within 3 months of the procedure
18. Subject has had a Cerebrovascular Accident (CVA) within 3 months of the procedure
19. Subject has a known allergy or intolerance to the device materials
20. Subject has a known allergy to anesthetic drugs
21. Subject has a known hypersensitivity or contraindication to anticoagulants, or contrast media, which is not amenable to pretreatment
22. Subject has active or systemic infection at the time of the index procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Verzini, Prof., Principal Investigator — A.O.U. Citta della Salute e della Scienza
Locations (16):
- Canada (2):
  - London Health Sciences Centre - Victoria Hospital, London
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec (IUCPQ), Québec
- Odense Universitetshospital, Odense, Denmark
- France (3):
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - CHU de Montpellier - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpitaux Universitaires de Strasbourg - Nouvel Hôpital Civil, Strasbourg
- Italy (5):
  - Policlinico Sant' Orsola - Malpighi, Bologna
  - IRCCS Ca' Granda Ospendale Maggiore Policlinico, Milan
  - Ospedale San Raffaele - Milano, Milan
  - Università di Perugia - Ospedale S.M. Della Misericordia, Perugia
  - IRCCS Policlinico San Donato, San Donato Milanese
- Netherlands (2):
  - Maastricht Universitair Medisch Centrum (MUMC), Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
- United Kingdom (3):
  - Cambridge University Hospitals NHS Foundation Trust - Addenbrooke's Hospital, Cambridge
  - Imperial College Healthcare NHS Trust - St Mary's Hospital, London
  - Saint George's Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verzini F, Cieri E, Kahlberg A, Sternbach Y, Heijmen R, Ouriel K, Robaina S, Azizzadeh A. A preliminary analysis of late structural failures of the Navion stent graft in the treatment of descending thoracic aortic aneurysms. J Vasc Surg. 2021 Oct;74(4):1125-1134.e2. doi: 10.1016/j.jvs.2021.04.018. Epub 2021 Apr 20. PMID 33892122
- [Derived] Azizzadeh A, Desai N, Arko FR 3rd, Panneton JM, Thaveau F, Hayes P, Dagenais F, Lei L, Verzini F. Pivotal results for the Valiant Navion stent graft system in the Valiant EVO global clinical trial. J Vasc Surg. 2019 Nov;70(5):1399-1408.e1. doi: 10.1016/j.jvs.2019.01.067. Epub 2019 May 21. PMID 31126765

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 subjects (53 US, 47 Outside US [OUS]), from 18 US sites and 15 OUS sites, contributed to the global cohort. The 1st subject was enrolled on 25 April 2016 (US) & on 08 June 2016 (OUS), the 100th subject on 28 March 2018.
Pre-assignment Details: A total of 152 subjects were consented to be reviewed for enrollment. 52 subjects were not approved for implantation, 100 subjects were approved for implantation. The 30-day primary endpoint was evaluated when 87 subjects completed 30-day follow-up.
Groups:
- Endovascular Repair: Subjects who were appropriate candidates for endovascular repair of Descending Thoracic Aortic Aneurysms (DTAA) and who met the inclusion and exclusion criteria.
Period: 30-Day Follow-up for Primary Endpoint
Arm/Group | Endovascular Repair
Started | 87 (The 30-day primary endpoint was evaluated when 87 subjects completed 30-day follow-up.)
Completed | 86
Not Completed | 1
Not completed — Death | 1
Period: 30-Day Follow-up for Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 100 (The 30-day secondary endpoint was evaluated when 100 subjects completed 30-day follow-up.)
Completed | 99
Not Completed | 1
Not completed — Death | 1
Period: 6-Month Follow-up Subject Accountability
Arm/Group | Endovascular Repair
Started | 99 (Note that 6-month follow up is not mandatory for OUS subjects)
Completed | 91
Not Completed | 8
Not completed — Death | 5
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1
Period: 12-Month Follow-up Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 91
Completed | 87
Not Completed | 4
Not completed — Death | 4
Period: 24-Month Follow-up Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 87
Completed | 52
Not Completed | 35
Not completed — Death | 2
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2
Not completed — Subject declined reconsenting to extended follow-up out to 5 years | 28
Period: 36-Month Follow-up Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 52
Completed | 48
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Period: 48-Month Follow-up Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 48
Completed | 42
Not Completed | 6
Not completed — Death | 4
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Period: 60-Month Follow-up Secondary Endpoint
Arm/Group | Endovascular Repair
Started | 42
Completed | 36
Not Completed | 6
Not completed — Death | 5
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Endovascular Repair: Subjects who were appropriate candidates for endovascular repair of Descending Thoracic Aortic Aneurysm (DTAA) and who met the inclusion and exclusion criteria. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 Outside US [OUS]).
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 60
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race data were not collected in OUS per regulation
  Participants
    number analyzed (Participants) | 53
    White | 42
    Non-White | 11
Region of Enrollment [Number; unit: participants]
  Canada | 7
  Netherlands | 4
  Denmark | 1
  United Kingdom | 8
  Italy | 17
  France | 10
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Composite Safety and Effectiveness Endpoint That is Based on the Percentage of Subjects Who Experienced (a) Access and/or Deployment Failures; and/or (b) Major Device Effect (MDE) Within 30 Days Post Index Procedure
Description: MDEs include: device-related secondary procedures, device-related mortality, conversion to open surgery, thoracic aortic aneurysm rupture.
  Access failure: Inability to insert device due to mechanical failure or anatomic exclusions of the femoral or iliac arteries.
  Deployment failure: Deployment failure due to subject anatomy or mechanical failure. Specifically, deployment of the stent graft from the delivery system.
  Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the primary endpoint global cohort of 87 subjects. The poolability on the primary endpoint between US and OUS data were assessed using Fisher's exact test.
Time Frame: 30 Days
Population: The 30-day primary endpoint was evaluated for Premarket Approval (PMA) when 87 subjects completed 30 day follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Repair: Valiant Evo Thoracic Stent Graft System: Procedure: thoracic endovascular aneurysm repair (TEVAR).
  Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the primary endpoint global cohort of 87 subjects (52 US, 35 OUS).
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 87
Participants | 2
Statistical Analysis 1: Comparison: Endovascular Repair; The primary study endpoint, major device effect at 30 days, is a dichotomous study outcome; hence, an exact method based on the binomial distribution was used for the hypothesis testing. The primary study endpoint was tested against a performance goal of 16%: H0: p ≥ 16% vs. Ha: p <16%, where p denotes the true event rate of primary study endpoint in the target population; Test type: Superiority; p < 0.0001, Exact binomial test; Event Rate = 0.023, 97.5% CI 1-sided [upper limit 0.081]

2. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety and Effectiveness outcome measures between 0-30 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 Outside US [OUS]).
  Measures include: peri-operative mortality, adverse events (AE), major adverse events (MAE), serious adverse events (SAE), secondary procedures, loss of stent graft patency, and endoleaks.
Time Frame: 30 Days
Population: Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 OUS).
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Repair: Subjects who were appropriate candidates for endovascular repair of Descending Thoracic Aortic Aneurysm and who met the inclusion and exclusion criteria. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 87 subjects (53 US, 47 OUS).
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  Peri-Operative Mortality | 2
  Adverse Events (AE) | 72
  Major Adverse Events (MAE) | 29
  Serious Adverse Events (SAE) | 32
  Secondary Procedures | 2
  Loss of Stent Graft Patency: number analyzed (Participants) | 95
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 94
  Endoleaks | 4

3. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety outcome measures between 0-183 days and Effectiveness outcome measures between 31-183 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort.
  Safety measures include: all-cause mortality (ACM), aneurysm related mortality (ARM), major device effects (MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE) and secondary procedures. Effectiveness measures include loss of stent graft patency, endoleaks, stent graft migration as compared to 1-month, and aneurysm expansion greater than 5 mm as compared to 1-month.
Time Frame: 6 Month
Population: Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International Trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 Outside US).
  Note that 6-month follow up is not mandatory for subjects enrolled under the Valiant Evo International protocol, resulting in fewer subjects analyzed at 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality (ACM): number analyzed (Participants) | 99
  All-Cause Mortality (ACM) | 6
  Aneurysm-Related Mortality (ARM): number analyzed (Participants) | 97
  Aneurysm-Related Mortality (ARM) | 3
  Major Device Effects (MDE): number analyzed (Participants) | 96
  Major Device Effects (MDE) | 2
  Adverse Events (AE) | 80
  Major Adverse Events (MAE) | 39
  Serious Adverse Events (SAE) | 50
  Secondary Procedures: number analyzed (Participants) | 96
  Secondary Procedures | 4
  Loss of Stent Graft Patency: number analyzed (Participants) | 53
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 52
  Endoleaks | 3
  Stent Graft Migration: number analyzed (Participants) | 55
  Stent Graft Migration | 0
  Aneurysm Expansion >5 mm relative to 1-Month: number analyzed (Participants) | 54
  Aneurysm Expansion >5 mm relative to 1-Month | 1

4. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety outcome measures between 0-365 days and Effectiveness outcome measures between 184-365 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort.
  Safety measures include: all-cause mortality (ACM), aneurysm related mortality (ARM), major device effects (MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE) and secondary procedures. Effectiveness measures include loss of stent graft patency, endoleaks, stent graft migration as compared to 1-month, and aneurysm expansion greater than 5 mm as compared to 1-month.
Time Frame: 12 Month
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Endovascular Repair: Subjects who were appropriate candidates for endovascular repair of Descending Thoracic Aortic Aneurysm and who met the inclusion and exclusion criteria. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 OUS).
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality (ACM): number analyzed (Participants) | 97
  All-Cause Mortality (ACM) | 10
  Aneurysm-Related Mortality (ARM): number analyzed (Participants) | 90
  Aneurysm-Related Mortality (ARM) | 3
  Major Device Effects (MDE): number analyzed (Participants) | 90
  Major Device Effects (MDE) | 4
  Adverse Events (AE) | 82
  Major Adverse Events (MAE) | 44
  Serious Adverse Events (SAE) | 55
  Secondary Procedures: number analyzed (Participants) | 89
  Secondary Procedures | 5
  Loss of Stent Graft Patency: number analyzed (Participants) | 79
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 78
  Endoleaks | 5
  Stent Graft Migration: number analyzed (Participants) | 79
  Stent Graft Migration | 0
  Aneurysm Expansion >5 mm relative to 1-Month: number analyzed (Participants) | 78
  Aneurysm Expansion >5 mm relative to 1-Month | 4

5. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety outcome measures between 0-730 days and Effectiveness outcome measures between 366-730 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort.
  Safety measures include: all-cause mortality (ACM), aneurysm related mortality (ARM), major device effects (MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE) and secondary procedures. Effectiveness measures include loss of stent graft patency, endoleaks, stent graft migration as compared to 1-month, and aneurysm expansion greater than 5 mm as compared to 1-month.
Time Frame: 24 Month
Population: Subjects who were appropriate candidates for endovascular repair of Descending Thoracic Aortic Aneurysm and who met the inclusion and exclusion criteria. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort of 100 subjects (53 US, 47 OUS).
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality (ACM): number analyzed (Participants) | 80
  All-Cause Mortality (ACM) | 13
  Aneurysm-Related Mortality (ARM): number analyzed (Participants) | 72
  Aneurysm-Related Mortality (ARM) | 3
  Major Device Effects (MDE): number analyzed (Participants) | 72
  Major Device Effects (MDE) | 5
  Adverse Event (AE): number analyzed (Participants) | 99
  Adverse Event (AE) | 85
  Major Adverse Event (MAE): number analyzed (Participants) | 99
  Major Adverse Event (MAE) | 49
  Serious Adverse Event (SAE): number analyzed (Participants) | 99
  Serious Adverse Event (SAE) | 62
  Secondary Procedures: number analyzed (Participants) | 71
  Secondary Procedures | 6
  Loss of Stent Graft Patency: number analyzed (Participants) | 52
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 50
  Endoleaks | 2
  Stent Graft Migration: number analyzed (Participants) | 51
  Stent Graft Migration | 0
  Aneurysm Expansion >5 mm relative to 1-Month: number analyzed (Participants) | 53
  Aneurysm Expansion >5 mm relative to 1-Month | 4

6. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety outcome measures between 0-1095 days and Effectiveness outcome measures between 731-1095 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort.
  Safety measures include: all-cause mortality (ACM), aneurysm related mortality (ARM), major device effects (MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE) and secondary procedures. Effectiveness measures include loss of stent graft patency, endoleaks, stent graft migration as compared to 1-month, and aneurysm expansion greater than 5 mm as compared to 1-month.
Time Frame: 36 Month
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality: number analyzed (Participants) | 78
  All-Cause Mortality | 14
  Aneurysm-Related Mortality: number analyzed (Participants) | 67
  Aneurysm-Related Mortality | 3
  Major Device Effects (MDE): number analyzed (Participants) | 68
  Major Device Effects (MDE) | 6
  Adverse Event (AE): number analyzed (Participants) | 99
  Adverse Event (AE) | 88
  Major Adverse Event (MAE): number analyzed (Participants) | 99
  Major Adverse Event (MAE) | 52
  Serious Adverse Event (SAE): number analyzed (Participants) | 99
  Serious Adverse Event (SAE) | 66
  Secondary Procedures: number analyzed (Participants) | 68
  Secondary Procedures | 6
  Loss of Stent Graft Patency: number analyzed (Participants) | 37
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 36
  Endoleaks | 3
  Stent Graft Migration: number analyzed (Participants) | 42
  Stent Graft Migration | 1
  Aneurysm Expansion >5mm relative to 1-Month: number analyzed (Participants) | 40
  Aneurysm Expansion >5mm relative to 1-Month | 4

7. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety outcome measures between 0-1460 days and Effectiveness outcome measures between 1096-1460 days post implant procedure. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort.
  Safety measures include: all-cause mortality (ACM), aneurysm related mortality (ARM), major device effects(MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE) and secondary procedures. Effectiveness measures include loss of stent graft patency, endoleaks, stent graft migration as compared to 1-month, and aneurysm expansion greater than 5 mm as compared to 1-month.
Time Frame: 48 month
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality (ACM): number analyzed (Participants) | 71
  All-Cause Mortality (ACM) | 20
  Aneurysm-Related Mortality (ARM): number analyzed (Participants) | 56
  Aneurysm-Related Mortality (ARM) | 4
  Major Device Effects (MDE): number analyzed (Participants) | 57
  Major Device Effects (MDE) | 8
  Adverse Events (AE): number analyzed (Participants) | 98
  Adverse Events (AE) | 90
  Major Adverse Events (MAE): number analyzed (Participants) | 98
  Major Adverse Events (MAE) | 55
  Serious Adverse Events (SAE): number analyzed (Participants) | 98
  Serious Adverse Events (SAE) | 69
  Secondary Procedures: number analyzed (Participants) | 57
  Secondary Procedures | 9
  Loss of Stent Graft Patency: number analyzed (Participants) | 42
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 40
  Endoleaks | 6
  Stent Graft Migration: number analyzed (Participants) | 45
  Stent Graft Migration | 2
  Aneurysm Expansion>5 mm relative to 1-Month: number analyzed (Participants) | 44
  Aneurysm Expansion>5 mm relative to 1-Month | 6

8. Secondary Outcome: Safety and Effectiveness Outcome
Description: Safety and Effectiveness outcome measures between implant procedure and 60 months. Data from the Valiant Evo US trial (NCT02652949) and Valiant Evo International trial (NCT02625324) were combined to create the global cohort. Measures include: aneurysm related mortality (ARM), major device effects (MDE), adverse events (AE), major adverse events (MAE), serious adverse events (SAE), secondary procedures, loss of stent graft patency, stent graft migration compared to 1 month imaging, aneurysm expansion greater than 5 mm compared to 1 month imaging, and endoleaks.
Time Frame: 60 Month
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Repair
Number analyzed (Participants) | 100
Participants
  All-Cause Mortality (ACM): number analyzed (Participants) | 66
  All-Cause Mortality (ACM) | 23
  Aneurysm-Related Mortality (ARM): number analyzed (Participants) | 48
  Aneurysm-Related Mortality (ARM) | 4
  Major Device Effects (MDE): number analyzed (Participants) | 49
  Major Device Effects (MDE) | 13
  Adverse Events (AE): number analyzed (Participants) | 97
  Adverse Events (AE) | 93
  Major Adverse Events (MAE): number analyzed (Participants) | 97
  Major Adverse Events (MAE) | 59
  Serious Adverse Events (SAE): number analyzed (Participants) | 97
  Serious Adverse Events (SAE) | 75
  Secondary Procedures: number analyzed (Participants) | 49
  Secondary Procedures | 14
  Loss of Stent Graft Patency: number analyzed (Participants) | 34
  Loss of Stent Graft Patency | 0
  Endoleaks: number analyzed (Participants) | 34
  Endoleaks | 8
  Stent Graft Migration: number analyzed (Participants) | 35
  Stent Graft Migration | 2
  Aneurysm Expansion >5 mm relative to 1-Month: number analyzed (Participants) | 34
  Aneurysm Expansion >5 mm relative to 1-Month | 5

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality at 30 Days, 6 Months, 12 Months, 24 Months, 36 Months, 48 Months, and 60 Months
Groups:
- Endovascular Repair 30-Day Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality, or one or more serious adverse event within 0-30 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 30-Day time period or were followed for at least 1 day.
  For Adverse Events, the 30-Day time period for reporting is 0-30 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 30-Day time interval.
- Endovascular Repair 6-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-183 days, or one or more serious adverse event within 31-183 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 6-Month time period or were followed for at least 91 days.
  For Adverse Events, the 6-Month time period for reporting is 31-183 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 6-Month time interval.
- Endovascular Repair 12-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-365 days, or one or more serious adverse event within 184-365 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 12-Month time period or were followed for at least 305 days.
  For Adverse Events, the 12-Month time period for reporting is 184-365 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 12-Month time interval.
- Endovascular Repair 24-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-730 days, or one or more serious adverse event within 366-730 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 24-Month time period or were followed for at least 549 days.
  For Adverse Events, the 24-Month time period for reporting is 366-730 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 24-Month time interval.
- Endovascular Repair 36-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-1095 days, or one or more serious adverse event within 731-1095 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 36-Month time period or were followed for at least 914 days.
  For Adverse Events, the 36-Month time period for reporting is 731-1095 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 36-Month time interval.
- Endovascular Repair 48-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-1460 days, or one or more serious adverse event within 1096-1460 days Procedure: thoracic endovascular aneurysm repair (TEVAR)
  For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 48-Month time period or were followed for at least 1279 days.
  For Adverse Events, the 48-Month time period for reporting is 1096-1460 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 48-Month time interval.
- Endovascular Repair 60-Month Secondary Endpoint: Subjects treated with the Valiant Evo Thoracic Stent Graft, who experienced all-cause mortality within 0-1825 days, or one or more serious adverse event within 1461-1825 days Procedure: thoracic endovascular aneurysm repair (TEVAR) For All-Cause Mortality, the number of participants at risk includes all enrolled subjects who either had an event within the 60-Month time period or were followed for at least 1644 days.
  For Adverse Events, the 60-Month time period for reporting is 1461-1825 days. The number of participants at risk includes the number of subjects at risk at the beginning of the 60-Month time interval.
Arm/Group | Endovascular Repair 30-Day Secondary Endpoint | Endovascular Repair 6-Month Secondary Endpoint | Endovascular Repair 12-Month Secondary Endpoint | Endovascular Repair 24-Month Secondary Endpoint | Endovascular Repair 36-Month Secondary Endpoint | Endovascular Repair 48-Month Secondary Endpoint | Endovascular Repair 60-Month Secondary Endpoint
All-Cause Mortality (participants affected / at risk) | 2/100 | 6/99 | 10/97 | 13/80 | 14/78 | 20/71 | 23/66
Serious Adverse Events (participants affected / at risk) | 32/100 | 27/98 | 22/91 | 17/84 | 14/66 | 17/62 | 15/49
Other Adverse Events (participants affected / at risk) | 62/100 | 32/98 | 20/91 | 21/84 | 14/66 | 16/62 | 14/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Repair 30-Day Secondary Endpoint (N=100) | Endovascular Repair 6-Month Secondary Endpoint (N=98) | Endovascular Repair 12-Month Secondary Endpoint (N=91) | Endovascular Repair 24-Month Secondary Endpoint (N=84) | Endovascular Repair 36-Month Secondary Endpoint (N=66) | Endovascular Repair 48-Month Secondary Endpoint (N=62) | Endovascular Repair 60-Month Secondary Endpoint (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anaemia Of Chronic Disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splenic lesion (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 2 | 1 | 1 | 0 | 0 | 0
Atrioventricular Block (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 1 | 1 | 2 | 1 | 0 | 0
Coronary Artery Dissection (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Coronary Artery Occlusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Node Dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal Incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Change of Bowel Habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fistula of Small Intestine (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Intestinal Strangulation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Small Intestine Obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Death (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Stent-Graft Endoleak (General disorders) | 1 | 1 | 0 | 0 | 1 | 3 | 3
Vascular Stent Thrombosis (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Anaphylactic Shock (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 5 | 2 | 0 | 1 | 1
Pulmonary Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 2 | 2 | 2 | 0 | 0 | 0 | 1
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Device Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incomplete Spinal Fusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative Delirium (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory Tract Procedural Complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Spinal Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tracheal Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Failure to Thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bladder Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intraductal Papillary Mucinous Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung Squamous Cell Carcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebellar Infarction (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 1 | 1
Dementia with Lewy Bodies (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolic Stroke (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Guillain-Barre Syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lacunar Stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolic Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Parkinson's Disease (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal Cord Ischaemia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vascular Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device Breakage (Product Issues) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Delirium Tremens (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 2
End Stage Renal Disease (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal Tubular Necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ureteric Obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Bladder Polyp (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 2 | 1 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 2 | 1 | 3 | 1 | 2 | 1
Aortic Dissection (Vascular disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Aortic Rupture (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atheroembolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertensive Urgency (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Iliac Artery Stenosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral Artery Occlusion (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral Artery Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Microcytic Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intervertebral Discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia Aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular Access Site Thrombosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug Withdrawal Convulsions (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Iliac Artery Dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Complication Associated With Device (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device Physical Property Issue (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive Emergency (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Artery Stenosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ischaemic Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Repair 30-Day Secondary Endpoint (N=100) | Endovascular Repair 6-Month Secondary Endpoint (N=98) | Endovascular Repair 12-Month Secondary Endpoint (N=91) | Endovascular Repair 24-Month Secondary Endpoint (N=84) | Endovascular Repair 36-Month Secondary Endpoint (N=66) | Endovascular Repair 48-Month Secondary Endpoint (N=62) | Endovascular Repair 60-Month Secondary Endpoint (N=49)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 1 | 0 | 0 | 0 | 0
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 5 | 2 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 0 | 0 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Valve Stenosis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 2 | 1 | 1 | 1 | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block First Degree (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 2 | 2 | 1 | 0 | 0 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypertensive Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus Tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Torsade De Pointes (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular Extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Congenital Hypercoagulation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Loeys-Dietz Syndrome (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Angiectasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presbyoesophagus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chest Pain (General disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0
Facial Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 0
Generalized Oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Non-Cardiac Chest Pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Swelling (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Puncture Site Haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 6 | 0 | 0 | 0 | 0 | 0 | 0
Stent-Graft Endoleak (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Central Nervous System Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epididymitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal Candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 1 | 0 | 1 | 1 | 0
Pneumonia Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post Procedural Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 3 | 1 | 3 | 0 | 1 | 1
Anaemia Postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aortic Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal Abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Incision Site Erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ligament Rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Post Procedural Fever (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Postimplantation Syndrome (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Postoperative Delirium (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative Respiratory Failure (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Hypotension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Site Reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sternal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular Access Site Complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Magnesium Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood Pressure Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine Output Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 0 | 0 | 0 | 1 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asterixis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Dissection (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0
Morton's Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neurological Decompensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parkinson's Disease (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radial Nerve Palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Cord Infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Spinal Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 1
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Focal Segmental Glomerulosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Renal Failure (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Renal Ischaemia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal Mass (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 3 | 0 | 1 | 0 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 2 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diaphragmatic Paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung Consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung Infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lung Opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Painful Respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 1 | 2 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Keloid Scar (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin Reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aortic Aneurysm (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 2 | 0
Aortic Dissection (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 7 | 4 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 4 | 1 | 0 | 0 | 0 | 0 | 0
Jugular Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Peripheral Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral Ischaemia (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Subclavian Artery Stenosis (Vascular disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0
Subclavian Artery Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial Septal Defect (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chondrodermatitis Nodularis Chronica Helicis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Visual Impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Injury Associated With Device (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Periorbital Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penetrating Aortic Ulcer (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penetrating Atherosclerotic Ulcer (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral Artery Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Angina Unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Congenital Aortic Valve Incompetence (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retroperitoneal Haematoma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Adverse Drug Reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Popliteal Pulse Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vocal Cord Paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bladder Hypertrophy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal Arteriosclerosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aortic Dilatation (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subclavian Artery Dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular Wall Hypertrophy (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Impaired Self Care (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal Nerve Palsy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Clinical evidence collected as part of the Valiant Evo US Clinical Trial (NCT02652949) and the Valiant Evo International Clinical Trial (NCT02625324) are combined to support commercial marketing approvals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medtronic owns the data of this clinical study, a single investigation site may access and use the data provided by itself for scientific publications following prior approval by Medtronic.

Pooling data from several investigation sites for publication purposes, national projects and international projects all require prior approval from Medtronic.

DOCUMENTS (2):
  • Study Protocol (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/24/NCT02625324/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT02625324/SAP_001.pdf